CLINICAL TRIAL: NCT00208728
Title: Prospective Evaluation of Modified Cardiopulmonary Bypass Circuits in the Pediatric Population
Brief Title: Cardiopulmonary Circuits in the Pediatric Population
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Brian Kogon, Principal Investigator, Emory University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0227-2003
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2013-11-27 (Estimated); Status verified 2013-11

CONDITIONS: Pediatric; Cardiac Surgery
Keywords: pediatric; congenital heart disease; cardiac surgery
MeSH Terms: conditions — Heart Defects, Congenital

INTERVENTIONS:
Device: PC/SMART cardiopulmonary bypass circuit
Device: PMEA modified cardiopulmonary bypass circuit
Device: Standard of care uncoated cardiopulmonary bypass circuit

SUMMARY:
During open-heart surgery, blood flow is supported by a heart-lung machine that both pumps the blood and gives it oxygen. A problem associated with a heart-lung machine is the damage to some of the blood caused by protein in the blood cell sticking to the sides of the heart-lung machine tubing. This breakdown of the blood cell affects the platelets, which help the blood to clot. Use of the un-treated circuit will be phased out within the next few years, as newer technology is available. The use of coated tubing has been shown to decrease problems with post-operative bleeding in the adult population. No studies have been done on the pediatric population. We plan to perform a prospective, randomized study using the un-treated circuits used now, the " Smart" circuit tubing manufactured by Cobe Cardiovascular Inc., Arvada, CO and the PMEA circuit manufactured by Terumo Corporation, Tokyo, Japan. Randomization will be performed by the perfusionist (the person that runs the heart-lung machine) in charge of the case. No one else will be aware of which circuit is being used. There will be no changes in the operation of the heart-lung machine, anesthesia or the surgery because of this study.

Blood testing that is standard of care and some additional tests will be performed on a small amount of blood drawn from. the patient via arterial lines. Additional blood sticks will not be required to obtain this sample.

DETAILED DESCRIPTION:
The goal of this study is to compare the PC/SMART and PMEA treated circuits against each other and the current clinical standard (untreated) circuit with regard to blood component damage during CPB.

Specific Aims SA1: To determine if the surface modified circuits decrease platelet activation, platelet sequestration, and fibrinolysis during pediatric cardiac surgery using CPB.

Hypothesis 1: Use of a surface modified circuit will attenuate the CPB related decrease in platelet count, diminish platelet dysfunction as measured by thromboelastography (TEG), and decrease fibrinolysis as measured by fibrin-split product levels and TEG.

SA2: To determine whether the use of surface modified circuits during pediatric cardiac surgery results in a clinically relevant decrease in post-operative coagulopathy as measured by post-operative bleeding and blood product use.

Hypothesis 2: The use of surface modified circuits will result in improved function of the coagulation system yielding less post-operative bleeding and thus fewer blood product transfusions.

Methods The study will be a prospective, randomized trial in which a total of 90 patients (5-10 kgs) undergoing first time cardiac surgery using CPB at Egleston Hospital will be randomized into 3 groups. Group 1 will be the control group for whom the current standard unmodified CPB circuit will be used. Group 2 will undergo surgery using the PC/SMART modified CPB circuit (Cobe Cardiovascular Inc, Arvada, CO). Group 3 will undergo surgery using the PMEA modified circuit (Terumo Corporation, Tokyo, Japan).

Hypothesis 1 will be tested using the following assays:

Total platelet count Hematocrit Prothrombin time (PT) Activated thromboplastin time (aPTT) Fibrin split-product level D-dimer level thromboglobulin level (ELISA assay) Thromboelastography (TEG) using heparinase (to eliminate heparin effect) both with and without REOPRO (a GPIIb/IIIa platelet inhibitor) to measure the relative contributions of platelet function and fibrinogen activity to clot formation

Performed at the following time-points:

T1 = after induction of anesthesia, prior to CPB T2 = 5 minutes after the initiation of CPB T3 = at the end of re-warming (end of CPB) T4 = post-bypass (five minutes after protamine administration) T5 = within 24 hours after surgery (TEG will not be collected at this time)

Hypothesis 2 will be tested by quantifying chest-tube drainage and blood product administration (red blood cells, platelets, fresh frozen plasma, and cryoprecipitate) over the first 12 hours after weaning off of CPB.

ELIGIBILITY:
Inclusion Criteria:

* patients electively scheduled for first time cardiac surgery requiring cardiopulmonary bypass
* weight between 5 kg and 10 kg
* signed informed consent

Exclusion Criteria:

* patients requiring emergent cardiac surgery
* patients who have undergone prior cardiothoracic surgery
* documented coagulation disorders
* use of anticoagulant drugs or anti-platelet agents within 48 hours of surgery
* patients who require more than 4 hours of CPB or require a return to CPB
* informed consent not obtained.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 90
Dates: Start 2003-05; Study Completion 2005-06

PRIMARY OUTCOMES:
Decrease in platelet activation, platelet sequestration and fibrinolysis.

SECONDARY OUTCOMES:
Decrease in post-operative coagulopathy as measured by bleeding and blood product use.

CONTACTS AND LOCATIONS:
Overall Officials: Paul Kirshbom, MD, Principal Investigator — Emory University and Children's Healthcare of Atlanta
Locations (1):
- Children's Healthcare of Atlanta, Atlanta, Georgia, United States

REFERENCES:
- [Background] Edmunds LH Jr. Blood-surface interactions during cardiopulmonary bypass. J Card Surg. 1993 May;8(3):404-10. doi: 10.1111/j.1540-8191.1993.tb00384.x. PMID 8507971
- [Background] Defraigne JO, Pincemail J, Dekoster G, Larbuisson R, Dujardin M, Blaffart F, David JL, Limet R. SMA circuits reduce platelet consumption and platelet factor release during cardiac surgery. Ann Thorac Surg. 2000 Dec;70(6):2075-81. doi: 10.1016/s0003-4975(00)01838-5. PMID 11156123
- [Background] Gunaydin S, Farsak B, Kocakulak M, Sari T, Yorgancioglu C, Zorlutuna Y. Clinical performance and biocompatibility of poly(2-methoxyethylacrylate)-coated extracorporeal circuits. Ann Thorac Surg. 2002 Sep;74(3):819-24. doi: 10.1016/s0003-4975(02)03796-7. PMID 12238845
- [Background] Gu YJ, Boonstra PW, Rijnsburger AA, Haan J, van Oeveren W. Cardiopulmonary bypass circuit treated with surface-modifying additives: a clinical evaluation of blood compatibility. Ann Thorac Surg. 1998 May;65(5):1342-7. doi: 10.1016/s0003-4975(98)00223-9. PMID 9594864
- [Background] Butler J, Rocker GM, Westaby S. Inflammatory response to cardiopulmonary bypass. Ann Thorac Surg. 1993 Feb;55(2):552-9. doi: 10.1016/0003-4975(93)91048-r. PMID 8431082